CLINICAL TRIAL: NCT01682681
Title: A Prospective, Observational, Multi-center Study to Assess Long-term Retention Rate of Topiramate in Patients With Epilepsy
Brief Title: An Observational Study to Evaluate Long-term Retention Rate of Topiramate in Participants With Epilepsy
Status: Completed | Type: Observational
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Other Study IDs: CR015865; TOPMATEPY4053
Record Dates: First submitted 2012-08-22; First posted 2012-09-11 (Estimated); Results first posted 2013-08-16 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-08

CONDITIONS: Epilepsy
Keywords: Epilepsy; Topiramate; Topmax
MeSH Terms: conditions — Epilepsy | interventions — Topiramate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Topiramate
  Interventions: Drug: Topiramate

INTERVENTIONS:
Drug: Topiramate — This is an observational study. Participants with seizures receiving topiramate as per Investigator's discretion will be observed.

SUMMARY:
The purpose of this study is to evaluate the long-term retention rate of topiramate in participants with epilepsy (seizure disorder).

DETAILED DESCRIPTION:
This is an open-label (a medical research study in which participants and researchers are told which treatments the participants are receiving, "unblinded"), single-arm, prospective (study following participants forward in time), observational (a clinical study in which participants identified as belonging to study groups are assessed for biomedical or health outcomes) and multi-center (when more than one hospital or medical school team work on a medical research study) study of topiramte in participants with epilesy. The study population will be all the epilepsy participants visiting outpatient study center over a period of two months. Topiramate will be administered as per Investigator's discretion for 52 weeks. Participants will visit the trial site for evaluation of endpoint at Baseline, Week 12, Week 26, and Week 52. Efficacy will primarily be evaluated by percentage of participants which will be retained to topiramate treatment uptil Week 52. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants with all type of epilepsy
* Participants with more than 2 episodes of seizure during last 1 year
* Participants who can comply with the visit schedule and are willing and able to complete evaluation procedures specified in the protocol during the treatment period
* Female participants with child bearing potential and who use proper contraceptive methods during the study period

Exclusion Criteria:

* Participants who have known hypersensitivity reaction or allergy to the study drug
* Participants who have taken topiramate within the three months of study start
* Participants who are determined not to be suitable for the clinical study participation by an Investigator's discretion
* Pregnant and nursing female participants

Ages: 2 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population will include participants with epilepsy who visit an out-patient clinic for two months and have not received topiramate treatment for at least three months prior to Screening.
Sampling Method: Non-Probability Sample
Enrollment: 1234 (Actual)
Dates: Start 2007-07; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Groups:
- Topiramate: This was an observational study. Participants with seizures received topiramate as per Investigator's discretion were observed.
Period: Overall Study
Arm/Group | Topiramate
Started | 1234
Treated | 1232 (2 Participants were not compliant with eligibility criteria)
Completed | 902
Not Completed | 332
Not completed — Lack of Efficacy | 62
Not completed — Withdrawal by Subject | 1
Not completed — Moved to other hospital | 10
Not completed — Lost to Follow-up | 174
Not completed — Adverse Event | 46
Not completed — tapering of topiramate | 5
Not completed — Other | 21
Not completed — Low compliance | 13

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS) population included all participants who met all the eligibility criteria.
Arm/Group | Topiramate
Number analyzed (Participants) | 1232
Age Continuous [Mean (Standard Deviation); unit: Years] | 24.07 (17.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 562
  Male | 670

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Retained to Topiramate Treatment
Description: Participants with long term retention of topiramate until 52 weeks were reported
Time Frame: Week 52
Population: The full analysis set (FAS) population included all participants who met all the eligibility criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 1232
Percentage of participants | 71.56 [68.95 to 73.99]

2. Secondary Outcome: Number of Participants Who Received Concomitant Antiepileptic Drugs (AEDs)
Description: Number of participants who received concomitant AEDs along with the topiramate were reported.
Time Frame: Baseline up to Week 52
Population: FAS population included all participants who met all the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Topiramate
Number analyzed (Participants) | 1232
Participants | 749

3. Secondary Outcome: Number of Participants Who Received Topiramate as First Mono-therapy, Second Mono-therapy or Add-on Therapy
Description: Number of participants who received topiramate as first mono-therapy (initial treatment of epilepsy with a single drug), second mono-therapy (second line treatment with a single drug) or add-on therapy (as a supplement therapy to another drug) were reported.
Time Frame: Baseline up to Week 52
Population: FAS population included all participants who met all the eligibility criteria.
Measure: Number; unit: Participants
Arm/Group | Topiramate
Number analyzed (Participants) | 1232
Participants
  First Mono-therapy | 507 (0)
  Second Mono-therapy | 64
  Add-on therapy | 661

4. Secondary Outcome: Percentage of Participants Without Seizure
Description: Participants without seizure was calculated as percentage of participants who were found to be free of seizures and were observed up to Week 52.
Time Frame: Baseline up to Week 52
Population: FAS population included all participants who met all the eligibility criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 1232
Percentage of participants | 40.50 [37.76 to 43.24]

5. Secondary Outcome: Percentage of Participants With Reduction in Seizure Frequency by 50 Percent or More
Description: Percentage of participants for whom seizure frequency was reduced by greater than or equal to 50 percent after topiramate treatment were reported.
Time Frame: Week 52
Population: FAS population included all participants who met all the eligibility criteria.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Topiramate
Number analyzed (Participants) | 1232
Percentage of participants | 84.20 [82.10 to 86.30]

ADVERSE EVENTS:
Time Frame: Baseline up to Week 52
Arm/Group | Topiramate
Serious Adverse Events (participants affected / at risk) | 8/1234
Other Adverse Events (participants affected / at risk) | 34/1234
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=1234)
Decreased appetite (Metabolism and nutrition disorders) | 1
Duodenal ulcer perforation (Gastrointestinal disorders) | 1
Hepatic neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Death (General disorders) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topiramate (N=1234)
Paraesthesia (Nervous system disorders) | 19
Weight decreased (Nervous system disorders) | 16

LIMITATIONS AND CAVEATS:
The study design is single arm and open label, so bias could not be excluded in the subjective evaluation by Participants and Investigators.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI cannot provide any trial related information to external parties' without mutual agreement with the Sponsor. This is valid even after the contract is canceled.